CLINICAL TRIAL: NCT05035979
Title: Oral Baidi Quzhi Granule Combined With Ju Ying Cream for Acne Vulgaris: Protocol for a Randomized, Double-blind, Multicenter Clinical Trial
Brief Title: Oral Baidi Quzhi Granule Combined With Ju Ying Cream for Acne Vulgaris
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai Skin Disease and Venereal Disease Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020045
Record Dates: First submitted 2020-06-13; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Randomized controlled trial; BaiDI QuZhi granule; Ju YIn cream; Traditional Chinese Medicine
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TCM comprehensive treatment group (Experimental): Participants in the TCM treatment group will receive BaiDi Quzhi granule two times daily after meals, Ju Yin cream therapy three times per week for 8 weeks.
  Interventions: Drug: BaidI Quzhi granule; Drug: Ju Yin cream
- TCM internal treatment group (Active Comparator): Participants in the TCM internal treatment group will receive Baidi Quzhi granule two times daily after meals and Ju Yin placebo therapy three times per week for 8 weeks.
  Interventions: Drug: BaidI Quzhi granule; Drug: Ju Yin placebo cream
- TCM external treatment group (Active Comparator): Participants in the TCM external treatment group will receive Baidi Quzhi placebo granule two times daily after meals and Ju Yin cream therapy three times per week for 8 weeks.
  Interventions: Drug: Ju Yin cream; Drug: Baidi Quzhi placebo granule
- Placebo group (Placebo Comparator): Participants in the placebo group will receive Baidi Quzhi placebo granule two times daily after meals, Ju Yin placebo therapy three times per week for 8 weeks.
  Interventions: Drug: Baidi Quzhi placebo granule; Drug: Ju Yin placebo cream

INTERVENTIONS:
Drug: BaidI Quzhi granule — Put each bag of medicine in one day into the same container, pour in about 50ml of warm water, stir until the granules are basically dissolved, add some boiled water to dilute, and take it twice.
  Other Names: Chinese Herbal Medicine
  Arms: TCM comprehensive treatment group; TCM internal treatment group
Drug: Ju Yin cream — Take JY cream 5g evenly applied to the face, negative ion spray at the same time acupoint massage along the meridian, apply 10min, clean the face with water, 3 times a week.
  Other Names: Chinese Herbal Medicine
  Arms: TCM comprehensive treatment group; TCM external treatment group
Drug: Baidi Quzhi placebo granule — Put each bag of medicine in one day into the same container, pour in about 50ml of warm water, stir until the granules are basically dissolved, add some boiled water to dilute, and take it twice.
  Other Names: Chinese Herbal Medicine
  Arms: Placebo group; TCM external treatment group
Drug: Ju Yin placebo cream — Take JY placebo cream 5g evenly applied to the face, negative ion spray at the same time acupoint massage along the meridian, apply 10min, clean the face with water, 3 times a week.
  Other Names: Chinese Herbal Medicine
  Arms: Placebo group; TCM internal treatment group

SUMMARY:
We designed the study as a double-blind,randomized,controlled clinical trial.The aim of this trial is to clarify the treatment efficacy, safety, and recurrence control of BaiDi QuZhi(BDQZ) granule combined with Ju Yin(JY) cream in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory skin disease of hair follicle and sebaceous gland, which is common in adolescents and adults.Systemic drugs commonly used in the treatment of acne include isotretinoin, oral antibiotics and hormone preparations. Isotretinoin is the first choice for the treatment of moderate and severe acne, but its use is limited by its adverse reactions such as cheilitis, elevated blood lipids and teratogenicity .The efficacy of BDQZ granule in the treatment of acne is accurate. However, large-scale randomized controlled trials have not been conducted on the efficacy, safety and recurrence of BDQZ granule. Therefore, our aim was to conduct a multicenter, randomized, double-blind, placebo-controlled clinical trial of oral BDQZ granule combined with JY cream in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with acne vulgaris aged from 16 to 45, male or female. 2. Patients who meet the western diagnostic criteria of mild and moderate acne vulgaris and the differentiation criteria of TCM syndrome (15,16).

3. Patients who voluntarily join this study with informed consent. 4. No acne drugs were received within 1 month, and no external drugs related to the disease were used within 1 week.

Exclusion Criteria:

* 1. Patients with severe primary diseases such as cerebrovascular, cardiovascular, liver, kidney and hematopoietic system.

  2. Participants will be ineligible if they ate pregnant or lactating women, and those with fertility plans in the next 2 years.

  3. Patients who do not meet the inclusion criteria, fail to use the medicine according to the regulations, fail to judge the curative effect, or incomplete data affect the judgment of curative effect or safety.

  4. Allergic constitution and allergic to the drug ingredients studied in this project.

  5. Cicatricial constitution. 6.Occupational acne caused by chemicals, acne caused by drugs.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 472 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of the investigators' overall assessment (IGA) for acne vulgaris | up to 16th weeks
  On the IGA (0-5) score, the percentage of subjects with IGA score reduction (baseline IGA- week 8 IGA) greater than or equal to 2 points.

SECONDARY OUTCOMES:
skin lesion count (total, inflammatory and non-inflammatory) | Patients will be evaluated at the 2st, 4nd, 6rd, 8th week and follow-up period (12th, 16th week).
  The change level of the investigators' overall assessment(IGA) score
Visual analogue scale (VAS) score of facial itching symptoms | Patients will be evaluated at the 2st, 4nd, 6rd, 8th week and follow-up period (12th, 16th week).
  VAS are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individiual patients and use this to achieve a rapid classification of symptom and disease control.
Visual analogue scale(VAS) score of facial pain symptoms | Patients will be evaluated at the 2st, 4nd, 6rd, 8th week and follow-up period (12th, 16th week).
  VAS are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individiual patients and use this to achieve a rapid classification of symptom and disease control.
Skindex-16 scale | Patients will be evaluated at the 2st, 4nd, 6rd, 8th week and follow-up period (12th, 16th week).
  A brief Quality-of-Life measure for patients with the skin diseases
Traditional Chinese Medicine(TCM) syndrome score | Patients will be evaluated at the 2st, 4nd, 6rd, 8th week and follow-up period (12th, 16th week).
  Score TCM syndromes such as tongue, pulse and clinical manifestations
Interleukin(IL)-17 | Patients will be evaluated at Baseline and at the 8th week.
  IL-17 was implicated in the pathogenic mechanisms of both inflammatory and infectious skin diseases such as staphylococcus infection, contact hypersensitivity, psoriasis and atopic dermatitis.
25-hydroxy Vitamin D | Patients will be evaluated at Baseline and at the 8th week.
  Vitamin D deficiency may have a role in the pathogenesis of acne
Dehydroepiandrosterone-sulfate(DHEA-S) | Patients will be evaluated at Baseline and at the 8th week.
  Adrenal steroid hormones produced by the secretion of the adrenal gland

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Shanghai Yueyang Intergrated Medicnie Hospital,Shanghai

IPD SHARING:
Plan to Share IPD: Undecided